CLINICAL TRIAL: NCT04683978
Title: Effect of Neck Extension on Intraocular Pressure in Patients Undergoing Palatoplasty
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, MD, Professor, Asan Medical Center
Other Study IDs: 2020-1854
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate | interventions — Patient Positioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Position — Neck extension

SUMMARY:
The purpose of this study is to investigate the change in intraocular pressure according to the neck extension during palatoplasty in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a palatoplasty with cleft palate and who are 6 months or older and under 24 months
* Patients with ASA class 1-2
* Patients who agree to voluntarily participate in this study

Exclusion Criteria:

* Patients who refused to participate in clinical studies
* History of diagnosis of neurologic or ophthalmic disease
* History of neurosurgery or ophthalmic surgery

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who have undergone a palatoplasty with cleft palate and who are 6 months or older and under 24 months
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure after neck extension | at 5 minutes after the position change (neck extension)
  Intraocular pressure after neck extension during palatoplasty

SECONDARY OUTCOMES:
Intraocular pressure 10 minutes after anesthetic induction | at 10 minutes after anesthetic induction (supine position)
  Intraocular pressure 10 minutes after anesthetic induction during palatoplasty
Intraocular pressure at end of surgery | immmediately after skin closure (neck extension)
  Intraocular pressure at end of surgery with neck extension
Intraocular pressure 5 minutes after supine position | at 5 minutes after the position change to the supine position (after the end of the surgery)
  Intraocular pressure 5 minutes after supine position

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yu J, Park JY, Jeong WS, Oh TS, Kim JY, Kim YK. Effect of neck extension on intraocular pressure in paediatric patients undergoing palatoplasty. J Plast Reconstr Aesthet Surg. 2023 Oct;85:309-315. doi: 10.1016/j.bjps.2023.07.014. Epub 2023 Jul 16. PMID 37541047